CLINICAL TRIAL: NCT02436564
Title: A Study Designed to Develop in Vitro Models of Liver, Biliary and Pancreatic Cancer for the Investigation of Tumour Biology and Potential Therapies
Brief Title: In Vitro Models of Liver and Pancreatic Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: The Gurdon Institute (Unknown); Ann McLaren Laboratory of Regenerative Medicine (Unknown)
Responsible Party: Principal Investigator, Dr. Kourosh Saeb-Parsy, University Lecturer and Consulatan Transplant Surgeon, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: A093484
Record Dates: First submitted 2015-04-30; First posted 2015-05-07 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Cholangiocarcinoma; Hepatocellular Carcinoma; Pancreatic Neoplasm
Keywords: pancreas; stem cells; tumours; in vitro models; organoids; cancer,; bile duct; liver
MeSH Terms: conditions — Cholangiocarcinoma; Carcinoma, Hepatocellular; Pancreatic Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — fresh tissue, frozen tissue
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: Organoid in vitro culture — Generation of 'organoids' using in vitro culture techniques, genomic DNA and RNA sequencing, application of genome editing technology, investigation of anti-tumour drugs, investigation of biological and functional properties of tumour cells, transplantation of organoid lines into animal models.

SUMMARY:
The primary objective is to develop an in vitro model of cancer for laboratory study using liver, biliary and pancreatic cancer tissue. The secondary objective is to study the genetic and cellular biology of cancer of the liver, biliary tract and the pancreas. As well the investigators hope to compare molecular and cellular biology of cancer cells with normal cells as well as potentially test the efficacy of current and future anti-cancer therapies.

Samples will be collected from tissue that has been resected as part of the treatment for a patient diagnosed with liver, bile duct or pancreas cancer.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients undergoing surgical resections for liver, biliary or pancreas cancers that are able to give informed consent.

Exclusion Criteria:

* Patients aged <18 or those who are unable to give informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are undergoing surgical resenctions of liver, biliary or pancreas cancers that are able to give informed consent
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2015-07; Primary Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Number of tumour-derived organoids successfully cultured in vitro for a minimum of 3 months. | 3 years

SECONDARY OUTCOMES:
Proportion of tumour-derived organoids that are genetically identical to the source tumour. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Kourosh Saeb-Parsy, PhD, FRCS, Principal Investigator — Cambridge Univeristy Hospitals
Locations (1):
- Addenbrooke's Hospital, Cambridge, United Kingdom